CLINICAL TRIAL: NCT01011647
Title: Prevalence of Sleep Disordered Breathing
Status: Terminated | Type: Observational
Why Stopped: Inadequate recruitment
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: 2042500
Record Dates: First submitted 2009-11-10; First posted 2009-11-11 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Unstable Angina; Acute Myocardial Infarction; Congestive Heart Failure
MeSH Terms: conditions — Angina, Unstable; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute coronary conditions: Patients hospitalized with the following conditions
  * Unstable angina
  * Acute myocardial infarction
  * Congestive heart failure

SUMMARY:
A novel technique in identifying unspecified sleep apnea has been developed. This technique uses signals typical acquired from a bedside monitor that is found in critical care environments. Those signals are then processed by a sleep analysis algorithm to provide an Apnoea Hypopnea Index (AHI) score. This study is intended to determine whether the prevalence of sleep disordered breathing identification among patients in a Coronary Care Unit (CCU) using this novel approach is significantly different than using routine techniques.

DETAILED DESCRIPTION:
This study will focus on inpatients diagnosed with coronary conditions. Specific eligibility criteria will include:

* Unstable angina
* Acute myocardial infarction
* Congestive heart failure Subjects enrolled in the study will be scored for sleep apnea using a novel approach designed by the sponsor. That score will not be used in the course of treatment. A follow-up call will determine whether the subject was identified for sleep disordered breathing during the hospital stay. A comparison will be done on the number of those identified with and without the use of the sleep scoring device.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or greater than 18 years at time of consent
* Written informed consent
* Patients admitted to the intensive care unit if able to remove oxygen
* Patients admitted to telemetry and step-down floor that will not require oxygen
* Primary diagnosis (any of the following)
* Un-stable angina
* Acute myocardial infarction
* Congestive heart failure

Exclusion Criteria:

* Previously diagnosed sleep disordered breathing
* Inability to consent
* Pregnancy
* Intubation (no longer excluded after extubation)
* Oxygen therapy (no longer excluded after therapy ends)
* End-Stage renal disease
* End-Stage liver disease
* Terminal disorders other than cardiac
* Severe scoliosis
* Cervical spinal cord injuries
* Neuromuscular disorders
* Severe COPD as defined by prescription of home oxygen therapy
* Other unsuitable circumstances

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject selection will come from patients admitted to the hospital with an acute cornonary condition.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2009-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Sleep disordered breathing was detected either by signals obtained from patient monitoring or by standard approaches by the site. | 3 months

SECONDARY OUTCOMES:
Length of CCU stay | 3 months
Length of hospital stay | 3 months
Prevalence of various sleep variables and correlation to known clinical and laboratory prognostic parameters | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- [Background] Guilleminault C, Tilkian A, Dement WC. The sleep apnea syndromes. Annu Rev Med. 1976;27:465-84. doi: 10.1146/annurev.me.27.020176.002341. No abstract available. PMID 180875
- [Background] Block AJ, Boysen PG, Wynne JW, Hunt LA. Sleep apnea, hypopnea and oxygen desaturation in normal subjects. A strong male predominance. N Engl J Med. 1979 Mar 8;300(10):513-7. doi: 10.1056/NEJM197903083001001. PMID 216912
- [Background] Sleep-related breathing disorders in adults: recommendations for syndrome definition and measurement techniques in clinical research. The Report of an American Academy of Sleep Medicine Task Force. Sleep. 1999 Aug 1;22(5):667-89. No abstract available. PMID 10450601
- [Background] Eckert DJ, Jordan AS, Merchia P, Malhotra A. Central sleep apnea: Pathophysiology and treatment. Chest. 2007 Feb;131(2):595-607. doi: 10.1378/chest.06.2287. PMID 17296668
- [Background] Young T, Palta M, Dempsey J, Skatrud J, Weber S, Badr S. The occurrence of sleep-disordered breathing among middle-aged adults. N Engl J Med. 1993 Apr 29;328(17):1230-5. doi: 10.1056/NEJM199304293281704. PMID 8464434
- [Background] Shamsuzzaman AS, Gersh BJ, Somers VK. Obstructive sleep apnea: implications for cardiac and vascular disease. JAMA. 2003 Oct 8;290(14):1906-14. doi: 10.1001/jama.290.14.1906. PMID 14532320
- [Background] Peters RW. Obstructive sleep apnea and cardiovascular disease. Chest. 2005 Jan;127(1):1-3. doi: 10.1378/chest.127.1.1. No abstract available. PMID 15653950
- [Background] Spurr KF, Graven MA, Gilbert RW. Prevalence of unspecified sleep apnea and the use of continuous positive airway pressure in hospitalized patients, 2004 National Hospital Discharge Survey. Sleep Breath. 2008 Aug;12(3):229-34. doi: 10.1007/s11325-007-0166-2. Epub 2008 Jan 31. PMID 18236092